CLINICAL TRIAL: NCT02460588
Title: Cyclophosphamide Added to Corticosteroid in the Treatment of Acute Exacerbation of Idiopathic Pulmonary Fibrosis: a Placebo-controlled Randomized Trial
Brief Title: Cyclophosphamide for Acute Exacerbation of Idiopathic Pulmonary Fibrosis
Acronym: EXAFIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P 140908; 2015-000492-27 (EudraCT Number)
Record Dates: First submitted 2015-03-16; First posted 2015-06-02 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Cyclophosphamide; Control Groups; Adrenal Cortex Hormones; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid with placebo (Placebo Comparator): Population is IPF patients with an AE who meet the inclusion and exclusion criteria defined below.
  All patients will receive non experimental medication with high dose of corticosteroid.
  Interventions: Drug: Placebo; Drug: Corticosteroid (prednisolone)
- Corticosteroid associated with Cyclophosphamide (Experimental): Population is IPF patients with an AE who meet the inclusion and exclusion criteria defined below.
  All patients will receive non experimental medication with high dose of corticosteroid.
  Intravenous Cyclophosphamide (CYC), 600 mg/m² (adapted to age and renal function, maximal dose of 1.2 g) at Day 0, Day 15, M1, M2
  Interventions: Drug: Cyclophosphamide; Drug: Corticosteroid (prednisolone)

INTERVENTIONS:
Drug: Cyclophosphamide — Population is IPF patients with an AE who meet the inclusion and exclusion criteria defined below.
  Intravenous Cyclophosphamide (CYC), 600 mg/m² (adapted to age and renal function, maximal dose of 1.2 g) at Day 0, Day 15, M1, M2
  Arms: Corticosteroid associated with Cyclophosphamide
Drug: Placebo — Population is IPF patients with an AE who meet the inclusion and exclusion criteria defined below.
  Other Names: Control group
  Arms: Corticosteroid with placebo
Drug: Corticosteroid (prednisolone) — All patients will receive non experimental medication with high dose of corticosteroid.
  Other Names: Both groups

SUMMARY:
Acute exacerbation of idiopathic pulmonary fibrosis (AE-IPF) is a major event of IPF with an annual incidence between 5 and 10% and is responsible for the death of one third of IPF patients. When AE-IPF occurs, it is associated with poor survival with an overall mortality at 3 months upper of 50%. To date, no treatment has been proved to be effective in AE-IPF but the efficacy of cyclophosphamide (CYC) on survival has been suggested, mainly by retrospective series and needs to be confirmed. This confirmation is mandatory to improve prognosis of AE-IPF but also to avoid unsuspected deleterious effect as it as been shown with immunosuppressor in stable IPF.

DETAILED DESCRIPTION:
Acute exacerbation of idiopathic pulmonary fibrosis (AE-IPF) is a major event of IPF with an annual incidence between 5 and 10% and is responsible for the death of one third of IPF patients. When AE-IPF occurs, it is associated with poor survival with an overall mortality at 3 months upper of 50%. To date, no treatment has been proved to be effective in AE-IPF but the efficacy of CYC on survival has been suggested, mainly by retrospective series and needs to be confirmed. This confirmation is mandatory to improve prognosis of AE-IPF but also to avoid unsuspected deleterious effect as it as been shown with immunosuppressor in stable IPF.

ELIGIBILITY:
Inclusion Criteria :

* ≥18 years of age
* Definite or probable IPF diagnosis defined on 2011 international recommendations
* Definite or suspicion of AE defined by IPFnet criteria after exclusion of alternative diagnosis of acute worsening.
* Efficient contraceptive method within 1 month for women and 3 months for men after the last dose of treatment
* Affiliation to the social security
* Able to understand and sign a written informed consent form

Exclusion Criteria:

* Identified etiology for acute worsening (i.e. infectious disease)
* Known hypersensitivity or contra-indication to CYC or to any component of the study treatment
* Patient on mechanical ventilation
* Active bacterial, viral, fungal or parasitic infection
* Active cancer
* Patient on a lung transplantation waiting list
* Treatment with CYC in the last 12 months
* Patient participating to another clinical trial
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
"Early" survival | 3 months
  All cause of mortality at 3 months

SECONDARY OUTCOMES:
Overall Survival | 6 months and 12 montns
  Overall Survival at M6 and M12
Respiratory disease-specific mortality | 6 months
  Respiratory disease-specific mortality at M3 and M6
Respiratory Morbidity | 6 months
  \Worsening dyspnea (0-100-mm visual analogue (VAS) scale anchored with 0 ''no breathlessness'' and 10 or 100 ''worst imaginable breathlessness". Worsening is defined an absolute decrease of 10 mm)
  * Or Increase need of supplemental oxygen of more than 3l/min to obtained a SaO2 > 90% or decrease of PaO2 of more than 10 mmHg with the same rate of flow supplemental oxygen
  * Or Decrease FVC of more than 10% of predicted value
  * Or Decrease diffuse capacity for carbon monoxide (DLCO) of more than 15% prednisolone
Chest HRCT features (HRCT images will be scored at 5 levels) | 6 months
  Chest HRCT features at M3 and M6 compared to inclusion
Prognosis factors of AE-IPF | 3 months
  PFTs results before AE-IPF
Time to visit after clinical worsening | 3 months
Laboratory evaluation (LDH, CRP) at AE diagnosis (composite) | 3 months
Prognosis factors of AE-IPF | 3 months
  PaO2 at AE diagnosis
Prognosis factors of AE-IPF | 3 months
  Chest HRCT features at AE diagnosis compared to HRCT before AE-IPF (if available)
Prognosis factors of AE-IPF | 3 months
  Chest HRCT classification before AE-IPF (definite UIP, probable UIP, indeterminate), if available
Time to dispense treatment of AE-IPF | 3 months
Hemorrhagic cystitis (occurence of hematuria on urine dipstick and pelvic pain and/or dysuria should lead to cystoscopy) | 6 months
Number of Infectious disease | 6 months
Diabetes mellitus (capillary blood glucose monitoring and fasting plasma glucose > 1.26 g/l) | 6 months
Hypertension (Blood pressure > 160/100 mmHg) | 6 months
Clinical laboratory evaluation (blood count, serum creatinin measurement composite) according to Common Terminology Criteria for Adverse Event (CTCAE). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc NACCACHE, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon, Paris, France

REFERENCES:
- [Background] Idiopathic Pulmonary Fibrosis Clinical Research Network; Raghu G, Anstrom KJ, King TE Jr, Lasky JA, Martinez FJ. Prednisone, azathioprine, and N-acetylcysteine for pulmonary fibrosis. N Engl J Med. 2012 May 24;366(21):1968-77. doi: 10.1056/NEJMoa1113354. Epub 2012 May 20. PMID 22607134
- [Background] Collard HR, Moore BB, Flaherty KR, Brown KK, Kaner RJ, King TE Jr, Lasky JA, Loyd JE, Noth I, Olman MA, Raghu G, Roman J, Ryu JH, Zisman DA, Hunninghake GW, Colby TV, Egan JJ, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kondoh Y, Lynch DA, Muller-Quernheim J, Myers JL, Nicholson AG, Selman M, Toews GB, Wells AU, Martinez FJ; Idiopathic Pulmonary Fibrosis Clinical Research Network Investigators. Acute exacerbations of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2007 Oct 1;176(7):636-43. doi: 10.1164/rccm.200703-463PP. Epub 2007 Jun 21. PMID 17585107
- [Background] Oishi K, Mimura-Kimura Y, Miyasho T, Aoe K, Ogata Y, Katayama H, Murata Y, Ueoka H, Matsumoto T, Mimura Y. Association between cytokine removal by polymyxin B hemoperfusion and improved pulmonary oxygenation in patients with acute exacerbation of idiopathic pulmonary fibrosis. Cytokine. 2013 Jan;61(1):84-9. doi: 10.1016/j.cyto.2012.08.032. Epub 2012 Sep 26. PMID 23021430
- [Background] Morawiec E, Tillie-Leblond I, Pansini V, Salleron J, Remy-Jardin M, Wallaert B. Exacerbations of idiopathic pulmonary fibrosis treated with corticosteroids and cyclophosphamide pulses. Eur Respir J. 2011 Dec;38(6):1487-9. doi: 10.1183/09031936.00127311. No abstract available. PMID 22130770
- [Background] Simon-Blancal V, Freynet O, Nunes H, Bouvry D, Naggara N, Brillet PY, Denis D, Cohen Y, Vincent F, Valeyre D, Naccache JM. Acute exacerbation of idiopathic pulmonary fibrosis: outcome and prognostic factors. Respiration. 2012;83(1):28-35. doi: 10.1159/000329891. Epub 2011 Aug 23. PMID 21860222
- [Background] Agarwal R, Jindal SK. Acute exacerbation of idiopathic pulmonary fibrosis: a systematic review. Eur J Intern Med. 2008 Jun;19(4):227-35. doi: 10.1016/j.ejim.2007.04.024. Epub 2008 Jan 16. PMID 18471669
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Cottin V, Crestani B, Valeyre D, Wallaert B, Cadranel J, Dalphin JC, Delaval P, Israel-Biet D, Kessler R, Reynaud-Gaubert M, Cordier JF, Aguilaniu B, Bouquillon B, Carre P, Danel C, Faivre JB, Ferreti G, Just N, Kouzan S, Lebargy F, Marchand Adam S, Philippe B, Prevot G, Stach B, Thivolet-Bejui F; French National Reference and Competence Centers for Rare Diseases; Societe de Pneumologies de Langue Francaise. [French practical guidelines for the diagnosis and management of idiopathic pulmonary fibrosis. From the National Reference and the Competence centers for rare diseases and the Societe de Pneumologie de Langue Francaise]. Rev Mal Respir. 2013 Dec;30(10):879-902. doi: 10.1016/j.rmr.2013.09.007. Epub 2013 Oct 25. No abstract available. French. PMID 24314711
- [Background] Nalysnyk L, Cid-Ruzafa J, Rotella P, Esser D. Incidence and prevalence of idiopathic pulmonary fibrosis: review of the literature. Eur Respir Rev. 2012 Dec 1;21(126):355-61. doi: 10.1183/09059180.00002512. PMID 23204124
- [Background] Wuyts WA, Agostini C, Antoniou KM, Bouros D, Chambers RC, Cottin V, Egan JJ, Lambrecht BN, Lories R, Parfrey H, Prasse A, Robalo-Cordeiro C, Verbeken E, Verschakelen JA, Wells AU, Verleden GM. The pathogenesis of pulmonary fibrosis: a moving target. Eur Respir J. 2013 May;41(5):1207-18. doi: 10.1183/09031936.00073012. Epub 2012 Oct 25. PMID 23100500
- [Background] Martinez FJ, Safrin S, Weycker D, Starko KM, Bradford WZ, King TE Jr, Flaherty KR, Schwartz DA, Noble PW, Raghu G, Brown KK; IPF Study Group. The clinical course of patients with idiopathic pulmonary fibrosis. Ann Intern Med. 2005 Jun 21;142(12 Pt 1):963-7. doi: 10.7326/0003-4819-142-12_part_1-200506210-00005. PMID 15968010
- [Background] Collard HR, Yow E, Richeldi L, Anstrom KJ, Glazer C; IPFnet investigators. Suspected acute exacerbation of idiopathic pulmonary fibrosis as an outcome measure in clinical trials. Respir Res. 2013 Jul 13;14(1):73. doi: 10.1186/1465-9921-14-73. PMID 23848435
- [Background] Churg A, Muller NL, Silva CI, Wright JL. Acute exacerbation (acute lung injury of unknown cause) in UIP and other forms of fibrotic interstitial pneumonias. Am J Surg Pathol. 2007 Feb;31(2):277-84. doi: 10.1097/01.pas.0000213341.70852.9d. PMID 17255773
- [Background] Papiris SA, Manali ED, Kolilekas L, Kagouridis K, Triantafillidou C, Tsangaris I, Roussos C. Clinical review: idiopathic pulmonary fibrosis acute exacerbations--unravelling Ariadne's thread. Crit Care. 2010;14(6):246. doi: 10.1186/cc9241. Epub 2010 Dec 22. PMID 21235829
- [Background] Song JW, Hong SB, Lim CM, Koh Y, Kim DS. Acute exacerbation of idiopathic pulmonary fibrosis: incidence, risk factors and outcome. Eur Respir J. 2011 Feb;37(2):356-63. doi: 10.1183/09031936.00159709. Epub 2010 Jul 1. PMID 20595144
- [Background] Akira M, Kozuka T, Yamamoto S, Sakatani M. Computed tomography findings in acute exacerbation of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2008 Aug 15;178(4):372-8. doi: 10.1164/rccm.200709-1365OC. Epub 2008 May 1. PMID 18451320
- [Background] Ambrosini V, Cancellieri A, Chilosi M, Zompatori M, Trisolini R, Saragoni L, Poletti V. Acute exacerbation of idiopathic pulmonary fibrosis: report of a series. Eur Respir J. 2003 Nov;22(5):821-6. doi: 10.1183/09031936.03.00022703. PMID 14621091
- [Background] Kim DS, Park JH, Park BK, Lee JS, Nicholson AG, Colby T. Acute exacerbation of idiopathic pulmonary fibrosis: frequency and clinical features. Eur Respir J. 2006 Jan;27(1):143-50. doi: 10.1183/09031936.06.00114004. PMID 16387947
- [Background] Fujimoto K, Taniguchi H, Johkoh T, Kondoh Y, Ichikado K, Sumikawa H, Ogura T, Kataoka K, Endo T, Kawaguchi A, Muller NL. Acute exacerbation of idiopathic pulmonary fibrosis: high-resolution CT scores predict mortality. Eur Radiol. 2012 Jan;22(1):83-92. doi: 10.1007/s00330-011-2211-6. Epub 2011 Aug 7. PMID 21822949
- [Background] Kondoh Y, Taniguchi H, Kitaichi M, Yokoi T, Johkoh T, Oishi T, Kimura T, Nishiyama O, Kato K, du Bois RM. Acute exacerbation of interstitial pneumonia following surgical lung biopsy. Respir Med. 2006 Oct;100(10):1753-9. doi: 10.1016/j.rmed.2006.02.002. Epub 2006 Apr 3. PMID 16584880
- [Background] Rice AJ, Wells AU, Bouros D, du Bois RM, Hansell DM, Polychronopoulos V, Vassilakis D, Kerr JR, Evans TW, Nicholson AG. Terminal diffuse alveolar damage in relation to interstitial pneumonias. An autopsy study. Am J Clin Pathol. 2003 May;119(5):709-14. doi: 10.1309/UVAR-MDY8-FE9F-JDKU. PMID 12760290
- [Background] Tomioka H, Sakurai T, Hashimoto K, Iwasaki H. Acute exacerbation of idiopathic pulmonary fibrosis: role of Chlamydophila pneumoniae infection. Respirology. 2007 Sep;12(5):700-6. doi: 10.1111/j.1440-1843.2007.01119.x. PMID 17875058
- [Background] de Groot K, Harper L, Jayne DR, Flores Suarez LF, Gregorini G, Gross WL, Luqmani R, Pusey CD, Rasmussen N, Sinico RA, Tesar V, Vanhille P, Westman K, Savage CO; EUVAS (European Vasculitis Study Group). Pulse versus daily oral cyclophosphamide for induction of remission in antineutrophil cytoplasmic antibody-associated vasculitis: a randomized trial. Ann Intern Med. 2009 May 19;150(10):670-80. doi: 10.7326/0003-4819-150-10-200905190-00004. PMID 19451574
- [Background] Tashkin DP, Elashoff R, Clements PJ, Goldin J, Roth MD, Furst DE, Arriola E, Silver R, Strange C, Bolster M, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel DE, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M; Scleroderma Lung Study Research Group. Cyclophosphamide versus placebo in scleroderma lung disease. N Engl J Med. 2006 Jun 22;354(25):2655-66. doi: 10.1056/NEJMoa055120. PMID 16790698
- [Background] Cottin V, Cadranel J, Crestani B, Dalphin JC, Delaval P, Israel-Biet D, Kessler R, Reynaud-Gaubert M, Valeyre D, Wallaert B, Bouquillon B, Cordier JF. Management of idiopathic pulmonary fibrosis in France: a survey of 1244 pulmonologists. Respir Med. 2014 Jan;108(1):195-202. doi: 10.1016/j.rmed.2013.11.017. Epub 2013 Dec 3. PMID 24361163
- [Result] Naccache JM, Jouneau S, Didier M, Borie R, Cachanado M, Bourdin A, Reynaud-Gaubert M, Bonniaud P, Israel-Biet D, Prevot G, Hirschi S, Lebargy F, Marchand-Adam S, Bautin N, Traclet J, Gomez E, Leroy S, Gagnadoux F, Riviere F, Bergot E, Gondouin A, Blanchard E, Parrot A, Blanc FX, Chabrol A, Dominique S, Gibelin A, Tazi A, Berard L, Brillet PY, Debray MP, Rousseau A, Kerjouan M, Freynet O, Dombret MC, Gamez AS, Nieves A, Beltramo G, Pastre J, Le Borgne-Krams A, Degot T, Launois C, Plantier L, Wemeau-Stervinou L, Cadranel J, Chenivesse C, Valeyre D, Crestani B, Cottin V, Simon T, Nunes H; EXAFIP investigators and the OrphaLung network. Cyclophosphamide added to glucocorticoids in acute exacerbation of idiopathic pulmonary fibrosis (EXAFIP): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2022 Jan;10(1):26-34. doi: 10.1016/S2213-2600(21)00354-4. Epub 2021 Sep 7. PMID 34506761
- [Derived] Naccache JM, Montil M, Cadranel J, Cachanado M, Cottin V, Crestani B, Valeyre D, Wallaert B, Simon T, Nunes H. Study protocol: exploring the efficacy of cyclophosphamide added to corticosteroids for treating acute exacerbation of idiopathic pulmonary fibrosis; a randomized double-blind, placebo-controlled, multi-center phase III trial (EXAFIP). BMC Pulm Med. 2019 Apr 11;19(1):75. doi: 10.1186/s12890-019-0830-x. PMID 30971235